CLINICAL TRIAL: NCT05115058
Title: A New Successful Approach for Emmetropic Presbyopic Patients Using Intrastromal Pocket With Smile Module
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EyeHP 1
Record Dates: First submitted 2021-11-05; First posted 2021-11-10 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: A New Successful Approach for Emmetropic Presbyopic Patients Using Intrastromal Pocket With Smile Module
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ReLex Smile module (Other): VisuMax femtosecond laser created the stromal pocket with a diameter 7.60 mm and cap thickness set to 120 μm from corneal surface and with a small opening - 2 mm superior incision at 90° and side cut angle 50°. The pocket was dissected using a blunt spatula.
  The patients were followed up for one year with distance, intermediate, and near visual acuity, slit lamp, corneal topography, anterior segment optical coherence tomography. Uncorrected near visual acuity at 35 cm increased from J7 to J2 in 8 eyes operated on, from J8 to J2 in 7 eyes, and from J6 to J2 in 6 eyes. Uncorrected intermediate visual acuity ranged from J4 to J5 at 70 cm, and uncorrected distance visual acuity remained binocular at 20/20. The patients reported satisfaction while reading a book, looking at the phone, and using a computer. No discomfort was observed from the lights while driving at night.
  Interventions: Other: relex Smile module

INTERVENTIONS:
Other: relex Smile module

SUMMARY:
Presbyopia is physiological insufficiency of accommodation associated with the aging of the eye that results in progressively worsening ability to focus clearly on close objects.Though presbyopia is a normal change in our eyes as we age, it often is a significant and emotional event because it's a sign of aging that's impossible to ignore and difficult to hide.

This defect is usually corrected by using glasses with bifocal power of suitable focal lengths.

But some patients don't want to use glasses for correction. In our study purpose is to show that near vision improves and patient satisfaction increases by preparing an intrastromal pocket for emmetropic patients with near vision problems using the SMILE module.

DETAILED DESCRIPTION:
This study started at 2016 was performed in Eye Hospital Pristina in 82 eyes of 41 patients aged (40-50) with the emmetropic presbyopic complaint.VisuMax femtosecond laser created the stromal pocket with a diameter 7.60 mm and cap thickness set to 120 μm from corneal surface and with a small opening - 2 mm superior incision at 90° and side cut angle 50°. The pocket was dissected using a blunt spatula.

The patients were followed up for one year with distance, intermediate, and near visual acuity, slit lamp, corneal topography, anterior segment optical coherence tomography. Uncorrected near visual acuity at 35 cm increased from J7 to J2 in 8 eyes operated on, from J8 to J2 in 7 eyes, and from J6 to J2 in 6 eyes. Uncorrected intermediate visual acuity ranged from J4 to J5 at 70 cm, and uncorrected distance visual acuity remained binocular at 20/20. The patients reported satisfaction while reading a book, looking at the phone, and using a computer. No discomfort was observed from the lights while driving at night. We are shaping the surface of the cornea via an introstrımal pocket. We are using the SMILE module without removing the lenticule, and we are just separating the center of the cap from the top of lenticule In the short term, we have observed increases in spherical aberrations of patients. We also think that corneal shaping has an effect on the presbyopic correction. We will see and analyze the long-term effects by observing them.

ELIGIBILITY:
Inclusion Criteria:

* patient not wishing to use glasses
* weak accomodation

Exclusion Criteria:

* active anterior segment pathology
* previous corneal or anterior segment surgery
* any infection

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Increase of near visual acuity | 12 months
  Preparing an intrastromal pocket for emmetropic patients with near vision problems using the SMILE module.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No